CLINICAL TRIAL: NCT05639114
Title: A Randomized, Double-blind, Parallel Group, Placebo-controlled Multicenter Phase 3 Study to Evaluate Efficacy, Safety and Tolerability of Two Regimens of Ianalumab on Top of Standard-of-care Therapy in Patients With Systemic Lupus Erythematosus (SIRIUS-SLE 1)
Brief Title: Phase 3 Study to Evaluate Two Regimens of Ianalumab on Top of Standard-of-care Therapy in Patients With Systemic Lupus Erythematosus (SIRIUS-SLE 1)
Acronym: SIRIUS-SLE 1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CVAY736F12301; 2022-002691-36 (EudraCT Number); 2023-508498-97-00 (Other: EU CT number)
Record Dates: First submitted 2022-11-04; First posted 2022-12-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; SLE; B cell depletion; SLEDAI-2K; BILAG-2004; SRI; ANA
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — ianalumab

STUDY DESIGN:
Intervention Model Description: The trial is designed to evaluate efficacy, safety and tolerability of two regimens of ianalumab compared to placebo, given as monthly or quarterly subcutaneous (s.c.) injection on top of standard-of-care (SoC) treatment in participants with active systemic lupus erythematosus (SLE).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Ianalumab s.c. monthly (Experimental): Ianalumab s.c. monthly
  Interventions: Drug: Ianalumab
- Ianalumab s.c. quarterly (Experimental): Ianalumab s.c. quarterly
  Interventions: Drug: Ianalumab
- Placebo s.c. monthly (Placebo Comparator): placebo s.c. monthly
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ianalumab — ianalumab s.c. monthly or quarterly
  Other Names: VAY736
  Arms: Ianalumab s.c. monthly; Ianalumab s.c. quarterly
Drug: Placebo — placebo s.c. monthly
  Arms: Placebo s.c. monthly

SUMMARY:
The trial will evaluate efficacy, safety and tolerability of two regimens of ianalumab compared to placebo, given as monthly or quarterly subcutaneous (s.c.) injection on top of standard-of-care (SoC) treatment in participants with active systemic lupus erythematosus (SLE).

DETAILED DESCRIPTION:
A randomized, double-blind, parallel group, placebo-controlled multicenter phase 3 study to evaluate efficacy, safety and tolerability of two regimens of ianalumab on top of standard-of-care therapy in patients with systemic lupus erythematosus (SIRIUS-SLE 1)

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 12 years or older at the time of screening, or limited to 18 years or older in European Economic Area countries and other countries where inclusion of participants below 18 years is not allowed.
* Diagnosis of systemic lupus erythematosus meeting the 2019 European League Against Rheumatism/American College of Rheumatology (EULAR/ACR) SLE classification criteria at least 6 months prior to screening.
* Elevated serum titers at screening of anti-nuclear antibodies ≥ 1:80 as determined by a central laboratory with a SLE-typical fluorescence pattern.
* Currently receiving CS and/or anti-malarial treatment and/or another disease-modifying antirheumatic drug (DMARD) as specified in the protocol.
* SLEDAI-2K criteria at screening: SLEDAI-2K score ≥ 6 points, excluding points attributed to "fever", "lupus headache", "alopecia", and "organic brain syndrome"
* BILAG-2004 disease activity level at screening of at least 1 of the following:

  * BILAG-2004 level 'A' disease in ≥ 1 organ system, Or
  * BILAG-2004 level 'B' disease in ≥ 2 organ systems
* Weigh at least 35 kg at screening

Exclusion Criteria:

* Prior treatment with ianalumab
* History of receiving following treatment: I) high dose CS, calcineurin inhibitors, JAK or other kinase inhibitors or other DMARD (except as listed in inclusion criteria) administered within 12 weeks prior to screening. II) cyclophosphamide or biologics such as immunoglobulins (intravenous or s.c.), plasmapheresis, anti-type I interferon receptor biologic agents, anti-CD40 agents, CTLA4-Fc Ig or B-cell activating factor (BAFF)-targeting agents administered within 24 weeks prior to screening; belimumab administered within 12 weeks prior to screening. III) any B cell-depleting therapies, other than ianalumab administered within 36 weeks prior to randomization or as long as B cell count is less than the lower limit of normal or baseline value prior to receipt of B cell-depleting therapy (whichever is lower). IV) Traditional Chinese medicines administered within 30 days prior to randomization.
* Active viral, bacterial or other infections requiring intravenous or intramuscular treatment for clinically significant infection
* Chronic infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Evidence of active tuberculosis infection
* History of primary or secondary immunodeficiency, including a positive human immunodeficiency virus (HIV) test result at screening
* Any one of the following abnormal laboratory values prior to randomization

  * Platelets < 25000/mm^3 (< 25 x 10^3/μL)
  * Hemoglobin (Hgb) < 8.0 g/dL (< 5 mmol/L), or < 7.0 g/dL (< 4.3 mmol/L) if related to participant's SLE such as in active hemolytic anaemia
  * Absolute neutrophil count (ANC) (< 0.8 x 10^3/ μL)
* Severe organ dysfunction or life-threatening disease at screening
* Presence of severe lupus kidney disease as defined by proteinuria above 2 g/day or equivalent using spot urine protein creatinine ratio, or serum creatinine greater than 2.0 mg/dL (176.84 µmol/L), or requiring immune-suppressive induction or maintenance treatment at screening
* Receipt of live/attenuated vaccine within a 4-week period before first dosing
* Any uncontrolled, co-existing serious disease, which in the opinion of the investigator will place the participant at risk for participation or interfere with evaluation for SLE-related symptoms
* Non-lupus conditions such as asthma, gout or urticaria, requiring intermittent or chronic treatment with systemic CS
* History of malignancy of any organ system other than localized basal cell carcinoma of the skin or in situ cervical cancer
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while on study treatment and for 6 months after stopping of investigational drug.
* Any surgical, medical, psychiatric or additional physical condition that may jeopardize participation in this study

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2023-03-02 (Actual); Primary Completion 2027-04-23 (Estimated); Study Completion 2029-04-20 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants on monthly ianalumab achieving Systemic Lupus Erythematosus Responder Index -4 (SRI-4) | Week 60
  SRI-4 response is defined as:
  * Systemic Lupus Erythematosus Disease Activity Index - 2000 (SLEDAI-2K) reduction from baseline of ≥ 4 points
  * No British Isles Lupus Assessment Group-2004 (BILAG-2004) worsening, defined as ≥ 1 new A or ≥ 2 new B items compared to baseline
  * No worsening in Physician Global Assessment of Disease Activity (PhGA), defined as an increase of ≥ 0.3 from baseline on a 0 to 3 visual analog scale

SECONDARY OUTCOMES:
Proportion of participants on monthly or quarterly ianalumab with no moderate or severe British Isles Lupus Assessment Group (BILAG) flare | Baseline to Week 60
  Moderate BILAG flare is defined as 2 or more new BILAG-2004 B items compared to the previous visit; severe BILAG flare is defined as (1 or more new BILAG-2004 A items compared to the previous visit)
Proportion of participants on monthly or quarterly ianalumab maintaining between Week 36 and Week 60 a reduced corticosteroid (CS) dose of predniso(lo)ne ≤ 5 mg/day or ≤ baseline dose, whichever is lower | Week 36 to Week 60
  Maintaining reduced CS dose from Week 36 to Week 60
Proportion of participants on monthly or quarterly ianalumab achieving BILAG-based Composite Lupus Assessment (BICLA) | Week 60
  BICLA response is defined as:
  * Reduction of all baseline BILAG-2004 A to B/C/D and baseline B to C/D and no worsening in other organ systems defined as ≥ 1 new A or ≥ 2 new B items compared to baseline
  * No worsening from baseline in SLEDAI-2K defined as an increase from baseline of > 0 points
  * No worsening in PhGA defined as an increase of ≥ 0.3 from baseline on a 0 to 3 PhGA visual analog scale
Proportion of participants on monthly or quarterly ianalumab achieving Lupus Low Disease Activity State (LLDAS) | Week 60
  LLDAS response is defined as:
  * SLEDAI-2K ≤ 4, with no activity in major organ systems (renal, central nervous system (CNS), cardiopulmonary, vasculitis, fever).
  * No new lupus disease activity compared with the previous assessment, defined as any new SLEDAI-2K component that was not present at the previous assessment
  * PhGA (scale 0-3) ≤ 1
  * Current predniso(lo)ne (or equivalent) dose ≤ 7.5 mg daily
  * Well tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents
Time to first occurrence of SRI-4 (participants on ianalumab monthly or quarterly) | Baseline to Week 60
  Time to first occurrence of SRI-4 from baseline to Week 60
Proportion of participants on monthly or quarterly ianalumab achieving SRI-4 at Week 60 while maintaining between Week 36 and Week 60 a reduced corticosteroid dose of predniso(lo)ne ≤ 5 mg/day or ≤ baseline dose, whichever is lower | Week 36 to Week 60
  Achieving SRI-4 at Week 60 while maintaining between Week 36 and Week 60 a reduced CS dose of predniso(lo)ne ≤ 5 mg/day or ≤ baseline dose, whichever is lower
Proportion of participants on monthly or quarterly ianalumab achieving SRI-6 | Week 60
  SRI-6 response is defined as:
  * SLEDAI-2K reduction from baseline of ≥ 6 points
  * No BILAG-2004 worsening, defined as ≥ 1 new A or ≥ 2 new B items compared to baseline
  * No worsening in PhGA, defined as an increase of ≥ 0.3 from baseline on a 0 to 3 visual analog scale
Proportion of participants on monthly or quarterly ianalumab achieving Short Form 36 (SF-36) Bodily Pain response | Week 60
  Achieving SF-36 Bodily Pain response
Proportion of participants on quarterly ianalumab achieving SRI-4 | Week 60
  SRI-4 response is defined as:
  * SLEDAI-2K reduction from baseline of ≥ 4 points
  * No BILAG-2004 worsening, defined as ≥ 1 new A or ≥ 2 new B items compared to baseline
  * No worsening in PhGA, defined as an increase of ≥ 0.3 from baseline on a 0 to 3 visual analog scale
Proportion of participants on monthly or quarterly ianalumab with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline to Week 60
  To evaluate safety and tolerability of ianalumab s.c. monthly or quarterly
Number of participants with adverse events | Baseline to Week 60
  To evaluate safety and tolerability of ianalumab s.c. monthly or quarterly
Proportion of participants with anti-ianalumab antibodies in serum (ADA assay) over time | Baseline to Week 164
  Immunogenicity of ianalumab s.c. monthly or quarterly
Ianalumab concentration in serum during the treatment and follow-up | Baseline to week 164
  Ianalumab concentration in serum

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (129):
- United States (29):
  - Pinnacle Research Group Llc, Anniston, Alabama
  - Providence Medical Center, Burbank, California
  - University of California San Diego, La Jolla, California
  - Keck School of Medicine, Los Angeles, California
  - Millennium Clinical Trials, Westlake Village, California
  - University of Colorado, Aurora, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - Clinical Res Of W Florida, Clearwater, Florida
  - GNP Research, Cooper City, Florida
  - University Of Miami, Miami, Florida
  - Clinical Research of West Florida Inc, Tampa, Florida
  - Parris and Associates Rheumatology, Lawrenceville, Georgia
  - Chicago Clinical Research Inst, Chicago, Illinois
  - Robert A Hozman MD SC, Skokie, Illinois
  - Lake Cumberland Rheumatology and In, New Albany, Indiana
  - Ochsner Clinic Foundation, Baton Rouge, Louisiana
  - Henry Ford Health, Detroit, Michigan
  - Univ of Nevada School of Med, Las Vegas, Nevada
  - Sahni Rheumatology and Therapy, West Long Branch, New Jersey
  - NYU Langone Health, Brooklyn, New York
  - Paramount Med Rsrch and Consult LLC, Middleburg Heights, Ohio
  - University Of Pittsburgh, Pittsburgh, Pennsylvania
  - Prisma Health, Columbia, South Carolina
  - Shelby Research LLC, Memphis, Tennessee
  - Accurate Clinical Research Research, Baytown, Texas
  - Novel Research LLC, Bellaire, Texas
  - Texas Arthritis Center, El Paso, Texas
  - Accurate Clinical Research, League City, Texas
  - Epic Medical Research, Red Oak, Texas
- Argentina (2):
  - Novartis Investigative Site, San Miguel, Tucumán Province
  - Novartis Investigative Site, San Miguel de Tucumán
- Brazil (11):
  - Novartis Investigative Site, Fortaleza, Ceará
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Belo Horizonte, Minas Gerais
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Recife, Pernambuco
  - Novartis Investigative Site, Niterói, Rio de Janeiro
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Salvador
- Bulgaria (3):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Rousse
  - Novartis Investigative Site, Sofia
- Canada (5):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Rimouski, Quebec
- China (17):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Haikou, Hainan
  - Novartis Investigative Site, Zhuzhou, Hunan
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Pingxiang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Linyi, Shandong
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Ningbo, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Xinxiang
- Colombia (3):
  - Novartis Investigative Site, Barranquilla, Atlántico
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Cali, Valle del Cauca Department
- Czechia (3):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Novartis Investigative Site, Guatemala City, Guatemala
- Hungary (4):
  - Novartis Investigative Site, Székesfehérvár, Fejér
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Zalaegerszeg
- Israel (2):
  - Novartis Investigative Site, Haifa
  - Novartis Investigative Site, Ramat Gan
- Japan (15):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa-ku
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Bunkyo-ku, Tokyo
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Fuchū, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Meguro City, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Miyazaki
  - Novartis Investigative Site, Osaka
- Poland (5):
  - Novartis Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Bytom
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Warsaw
- Portugal (3):
  - Novartis Investigative Site, Braga
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Vila Nova de Gaia
- Slovakia (2):
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Košice
- South Africa (4):
  - Novartis Investigative Site, Pretoria, Gauteng
  - Novartis Investigative Site, Cape Town, Western Cape
  - Novartis Investigative Site, Stellenbosch, Western Cape
  - Novartis Investigative Site, Umhlanga
- Spain (13):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Elche, Alicante
  - Novartis Investigative Site, Badalona, Barcelona
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, San Sebastian Reyes, Madrid
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
  - Novartis Investigative Site, Valladolid
- Thailand (3):
  - Novartis Investigative Site, Songkhla, Hat Yai
  - Novartis Investigative Site, Muang, Thailand
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Ankara, Bilkent Cankaya
  - Novartis Investigative Site, Ankara, Etlik
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Istanbul, Umraniye

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com